CLINICAL TRIAL: NCT03244215
Title: Evaluation Of Risk Of Recurrence Of Stroke And Vascular Events In Patients Presenting With Acute Stroke And Tia To Hamad General Hospital
Brief Title: The Recurrence Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr.Naveed Akhtar, Consultant Neurologist, Hamad Medical Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15304/15
Record Dates: First submitted 2017-06-04; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Acute Stroke; Transient Ischemic Attack
Keywords: Recurrence of stroke; Corneal Confocal Microscopy; High performance liquid chromatography,; Inflammatory biomarkers; modified Rankin scale ( mRS)
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): The intervention to be evaluated is the patient response and compliance to best medical treatment and prevention of recognized stroke risk factors and the recurrence of stroke and TIA in the study group and its relation to the incidence of blood biomarkers.
  The Nurse practitioners at the stroke ward will withdraw blood and collect urine samples from all the subjects. All the subjects from the study group will have 2 follow up visits (1 month and at 1 year) at HGH and one telephonic follow up at 3 months. The blood samples will be used to monitor blood inflammatory biomarker levels. At the beginning of the study, all subjects will have an MRI scan to assess plaque volume (this MRI scan will be ordered as part of the standard of care as per the policies applied to all stroke patients). MRI scans will be repeated at one year to assess any progression or regression in the plaque volume of the subjects.
  No drugs will be administered to the patients for the purpose of our study.
  Interventions: Diagnostic Test: Corneal Confocal Imaging; Diagnostic Test: Magnetic resonance Imaging; Other: Blood sample
- Control (Other): The control group will have blood work done to assess their blood inflammatory biomarkers but not the corneal confocal imaging.
  Interventions: Other: Blood sample

INTERVENTIONS:
Diagnostic Test: Corneal Confocal Imaging — Retinal imaging will be ordered for all subjects in the study group. Corneal
  Arms: The study group
Diagnostic Test: Magnetic resonance Imaging — MRI will be ordered for all study subjects at the completion of their participation at year 1. The MRI will assess the the progression or regression of the cerebrovascular health of the study subjects.
  Arms: The study group
Other: Blood sample — Blood samples will be obtained to evaluate the levels of blood inflammatory biomarkers in both the subjects and control group.

SUMMARY:
The primarily goal of the research is to better understand progression of disease in patients who present with an acute stroke to the Hamad General Hospital (HGH) stroke and Transient Ischemic Attack (TIA) clinic. The investigators are specifically interested in patients who have diabetes and have a stroke.

The patients enrolled into the research will have detailed clinical evaluation and their imaging studies (MRI and Doppler) will be reviewed. After informed consent, subjects will be examined in the stroke Ward /TIA clinic upon recruitment, and later at less than 48 hours of recruitment (blood extraction and urine samples) and for follow up visits at 1 month+/-7 days (clinical evaluation and to extract blood and urine samples), at 3 months (telephonic conversation only) and at 1 year (clinical and repeat MRI brain).

During the initial visit at the ward the investigators will collect serum and plasma for proteomic and metabolomic studies. These will be repeated at less than 48 hours and at 1 month+/-7 days. Investigators will test the effects of risk factors such as diabetes/stroke on the endothelial procoagulant and inflammatory state at onset and evaluate if best medical control leads to improvement in such markers.The repeated studies will determine if better management and presence of certain blood biomarkers can predict or translate to slower progression of disease and correlate it with clinical status.

DETAILED DESCRIPTION:
Patient admitted to the stroke service with acute stroke and TIAs will be eligible for the study. The study will enroll patients at Hamad General Hospital in the setting of the Stroke Ward.

The investigators anticipate approximately 300 patients to be enrolled based on the number of strokes that are admitted to the HGH stroke service every year.

The research primarily involves the evaluation of best medical therapy, and the incidence of biomarkers in the recurrence and progression of the disease in a high-risk cohort of stroke and TIA patients.

After obtaining informed consent the subjects medical information such as medical history will be collected in the case record forms. subjects MRI studies ( performed as standard of care) will be analyzed with a special software to determine the extent and volume of the most recent infarction. The degree of previous white matter damage and any incidental previous strokes will be recorded. MRI brain is a routine imaging technique in the care of stroke patients. Corneal confocal microscopy (CCM) imaging will be ordered for subjects whose standard of care attending physicians havent ordered for them. Some Stroke patients at HGH are ordered CCM if considered necessary by their physician. For the purpose of the study, the investigators would like to order CCM for all the subjects. CCM can be perfomed at anytime within the first month of recruitment into the study so the investigators will have it scheduled as it is convenient to the subjects within the month. The investigators hypothesize that corneal nerve loss may be driven by the same common vascular risk factors which may lead to stroke and thereby provide a surrogate for cerebral neuronal loss and hence pre-stroke 'neuronal reserve'. Hence CCM may allow us to identify the extent of risk factor burden. Furthermore, the quantification of corneal nerves may allow the identification of those with a lower pre-stroke neuronal reserve, and hence may suffer worse neurological outcomes following a stroke.

The subjects will be offered the best medical treatment for stroke, risk factors will be assessed by a team of stroke neurologists and nurse specialists. There will be regular follow-up visits at 1 month+/- 7 days, 3 months ( telephonic follow up only) and 1 year (clinical and repeat MRI brain).

After consent, serum and plasma will be obtained at onset of participation: Sample A (at onset), Sample B: within less than 48 hours, and Sample C:at 30 day +/- 1 week follow up visit. The blood samples will assist the team to study pro-coagulant and inflammatory markers. The team will require 10 mL ( 3 vials, 2 of which will have 4 mL of blood and the 3rd will have 2 mL) of blood on the aforementioned three days.

The blood , plasma and urine samples will undergo testing at the Neuroscience lab at iTRI, HMC, Qatar. A comparison between the different circulating biomarkers, proteins, DNA and metabolites might provide useful information on correlation between diabetes ( and other risk factors) and stroke. A variety of techniques are to be used including the following

1. Metabolites (metabolomics) High performance liquid chromatography (HPLC) and Liquid chromatography mass spectroscopy (LC/MS/MS) for detection of branching amino acids, glycine, aromatic amino acids and neurotransmitters.

   Molecular biology techniques for detection of cytokines and interleukins Measurement of microparticles and their content in human serum via flow cytometry ELISA for detection of reactive oxygen species SDS-PAGE for detection of cysteine proteases and inflammatory response proteins vWF testing to be done in Hamad General Hospital laboratory
2. Proteomics In the proposed study, th einvestigators will use a proteomics based approach to perform a global proteomic profiling using the plasma from patients reportedly suffering from ischemic stroke and are at the same time diabetic. The proteomic profiling could lead to the identification of set of novel proteins that can be used as potential markers involved in the ischemic stroke development in patients with diabetic condition. By using a gel-based proteomics approach, the plasma proteins will be subjected to pre-fractionation by SDS-PAGE analysis followed by in-gel tryptic digestion and the purified peptides will be analyzed by Liquid Chromatography coupled to tandem Mass Spectrometry. The sequenced peptides will be searched against the available database to obtain protein identifications.

Samples required: Serum, plasma and urine samples. Plasma can be retrieved from whole blood in EDTA sample bottles after centrifugation. Serum can be retrieved from whole blood in plain sample bottles after centrifugation. Urine can be collected in plain sample bacti bottles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years and older
* Subjects willing to give consent and agree to regular follow up visits;
* Male/Female patients of all nationalities admitted to HGH or seen in the Stroke Ward/ TIA clinics with a confirmed diagnosis of acute stroke and TIA, confirmed on the initial standard of care ordered MRI imaging.
* Stroke onset is less than 48 hours.

Exclusion Criteria:

* Pregnant women or individuals with cognitive disabilities.
* individuals with onset > 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2018-02-17 (Estimated); Study Completion 2018-05-17 (Estimated)

PRIMARY OUTCOMES:
Circulating Biomarkers | Blood samples will be assessed at baseline
  The primary outcome will be to assess blood inflammatory biomarker levels in both the study group as well as the controls at baseline
Circulating biomarkers | Blood samples will be extracted at 48 hours
  To assess blood inflammatory biomarker levels in the study group at less than 48 hours
Circulating biomarkers | Blood samples will be extracted at 1 month+/- 7 days
  To assess blood inflammatory biomarker levels in the study group at less than 1 month+/- 7 days

SECONDARY OUTCOMES:
Progression of disease | 1 year
  We will measure the plaque volume in the stroke patients by conducting an MRI scan at admission to the hospital and later repeating it at year 1. We will also utilize corneal confocal imaging as a surrogate procedure to assess the progression of stroke and other vascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Akhtar, MD, Principal Investigator — Hamad Medical Corporation; Ashfaq Shuaib, FRCPC, Study Chair — University of Alberta
Locations (1):
- The Neuroscience Institute, Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
We do not plan to share any IPD with other investigators.